CLINICAL TRIAL: NCT00938561
Title: Validity and Reliability of a Novel GFR Marker
Brief Title: Evaluation of New Markers to Assess Kidney Function
Status: Withdrawn | Type: Observational
Why Stopped: Non availability of funding
Sponsor: Tufts Medical Center (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 8608; 2008-08
Record Dates: First submitted 2009-07-08; First posted 2009-07-14 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Glomerular Filtration Rate; Kidney function; Markers
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Inulin

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Blood and urine will be retained for future testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- With and without Chronic Kidney Disease: A cohort of 10 patients subjects with and without kidney disease exhibiting a broad range of age and kidney function
  Interventions: Drug: Inulin

INTERVENTIONS:
Drug: Inulin

SUMMARY:
Glomerular filtration rate (GFR) is widely accepted as the best index of kidney function in health and disease, and accurate values are required for optimal clinical decision making and in large-scale epidemiologic studies and clinical trials. Current recommended methods for measuring GFR are expensive, cumbersome to administer and assay and requires urine collection and administration of radioactive materials. The purpose of this study is to evaluate two non-radioactive markers (iohexol and gadolinium) compared to urinary clearance of inulin and iothalamate. The investigators hypothesize that plasma clearance of non-radioactive markers will be unbiased compared to a gold standard and more precise than currently used urinary clearance methods.

DETAILED DESCRIPTION:
General description: The overall study procedure requires assessment of eligibility and safety for inclusion in the study through a) the screening questionnaire; b) medical history, which will be derived from subject and combined with a review of his/her medical record after signing the consent; and c) interview, physical examination and laboratory tests from screening visit if required.

Screening questionnaire: All subjects, whether they are interviewed during a clinic visit or call in response to fliers, will be given the pre-screening questionnaire. This will be given to people who voluntarily express interest in the study. Participants who do not disclose any conditions that would exclude them from participating will be invited to a health screening visit.

Health screening visit: The purpose of the pre-study health screening is to perform a more detailed assessment than is provided in the screening questionnaire to determine if potential subjects are eligible to participate in the study. A member of the research team will first read the consent form with the subject, describe the health screening and study visits, and answer any questions that the subject has regarding the nature of the study and/or study procedures. The screening visit will consist of the following:

* Reading and signing the study consent. The subject will be given a copy of the consent.
* Collection of information on demographics and current and past health history.
* Ascertain participants medical history through participant interview and a review of his/her medical record
* A physical exam, which will include measuring and recording vital signs (temperature, blood pressure, heart rate, breathing rate), height, weight (if not documented in medical record in past 3 months).
* Collection of a blood sample for laboratory testing, if required.
* Pre-menopausal women of child-bearing potential we will undergo a serum pregnancy test, using a small amount of blood from the sample collected above.
* Ascertainment of current and recent past medications.

If the subject is a patient at Tufts Medical Center, a research team member may access the potential participant's medical record after the subject has signed the consent form to further screen for potential exclusion criteria, ascertain laboratory test results that are necessary for determining eligibility, and confirm the medical history provided by the potential participant and medication list. If the participant is not a patient at Tufts Medical Center, then the research team member will obtain permission to obtain the participant's medical record from his/her physician.

For non-pregnant women of childbearing age (pre-menopausal) who are sexually active, use of an acceptable birth control method will be required for participation. They will be requested to sign a statement of compliance prior to participating in the study stating that they are employing one of the below-listed forms of contraception between the screening and study visits.

* condoms with spermicide
* diaphragm with spermicide
* injectable contraceptives (Depoprovera)
* transdermal contraceptives (Ortho-Evra and Nuvaring)
* intrauterine device (IUD)
* permanent sterilization (i.e. tubal ligation, vasectomy, essure)
* abstinence from sexual activity
* hysterectomy
* oral contraceptives

If the study visit occurs 3 weeks or more after the health screening, the female subjects will undergo a second, urine-based pregnancy test on the morning of the study visit. In addition, healthy women will be required to continue employing an accepted birth control method and not attempt to become pregnant for at least one month following completion of the final study visit. Women with CKD will be requested to continue employing an accepted birth control method for at least two months following completion of the final study visit.

If a potential subject is taking trimethoprim containing medications or cimetidine, the study physician will discuss with the attending physician whether it is safe for the person to stop these medications for one week prior to the study. If not, then the person will be excluded from participation. If a potential subject is taking non-steroidal anti-inflammatory agents or medications that block the renin-angiotensin system, the study physician will discuss with the potential participant and the attending physician whether maintenance of stable dose of these medications is possible. If a change in the subject's medication regimen is required immediately prior to the study visit, the subject will be rescheduled for a later date.

Eligibility will be determined by the principal investigator or other physician co-investigators based on the medical history obtained from the participant, and their medical records and the results of the laboratory test that were included in the medical record or obtained during the health screening visit). Eligible subjects will be contacted to see if they remain interested in participating in the study. A study visit date will then be scheduled. All subjects will receive a stipend for the health screening.

Screening prior to at-home dosing of KI The main concern when subjects are asked to take KI on the morning prior to the study visit is the possibility that the patient is allergic to iodine and will thus have a reaction to the KI in the unobserved environment at home. The research team will identify subjects with known allergies in advance by screening the subjects' medical records (if available) and through the health-history interview conducted via telephone by the study coordinator. Subjects who are not sure if they have an iodine allergy because they have not eaten shellfish or have never received contrast dye and, therefore, cannot say with sureness that they are not allergic will be excluded from participation.

Supplying the KI tablet to the subject prior to the study visit The KI tablet will be supplied to the study participant from 2 days to approximately 2 weeks prior to the study visit. The tablet and the instruction sheet will be mailed to the subject or supplied during the health screening visit at the Clinical and Translational Research Center (CTRC); however, if the subject is a patient at the KBPC and has an appointment with their physician within approximately 2 weeks of the study visit, a member of the research team may provide the KI tablet and instruction sheet at the clinic visit. Otherwise, all subjects will be asked to provide their mailing address during the phone interview to ensure that the tablet is sent to the correct address.

Per the IosatTM package insert, the tablet should be stored in a dry place at room temperature and out of direct sunlight. Subjects will also be instructed to keep the tablet in a place where someone else cannot accidentally consume it (i.e., a child, spouse, etc). These storage techniques will be conveyed to the subject in the included instructions. The tablets are available individually wrapped in foil blister packs to protect them from the effects of UV light, which can damage the KI. To further decrease the likelihood of damage to the tablet due to improper storage or handling, all tablets will be packaged in a secondary pill bottle with child-safe caps by the Tufts Medical Center pharmacy.

Subjects will be instructed to take the KI tablet on the morning of the day before the study visit between 6:00 AM and 10:00 AM. Instructions with the tablet will include:

* An additional warning, in bold typeface, instructing the subject to not take the tablet if they even suspect that they might have an iodine allergy.
* Proper administration. Per the package insert, the tablet can be consumed with water, low fat milk, low fat chocolate milk, or orange juice.
* Symptoms of an allergic reaction and steps to take in the event that the subject experiences a reaction (per the IosatTM package insert).

In addition to listing the emergency phone number '911' on the package, the contact numbers of Dr. Stevens (PI) and the study coordinator will be included in the event that the subject has any questions or concerns. On the morning of the study visit, the research staff will ask the subject to give verbal confirmation that they have taken the KI dose and record the approximate time at which the subject took it.

Subjects taking medications that interfere with creatinine, who can safely cease taking the medication, as described in the exclusion criteria, will be reminded to stop these medications 1 week prior to the study visit at this time. In addition, a member of the research team will contact the subject 2-3 days prior to the visit date to ensure that the subject is clear on all directions and has no questions or concerns. During this call, the subject will be reminded to take the KI tablet at the specified time. When possible, the study personnel will also call the subject at approximately 9:00 AM on the morning of the day before the study visit to ensure that the subject took the tablet.

Non-diabetic subjects will be requested to fast overnight and to avoid changes in non-steroidal anti-inflammatory agents or medications that block the renin-angiotensin system. Subjects with diabetes will be asked to eat a light breakfast the morning of the study visit. Subjects will be asked to maintain adequate oral hydration and to ingest two to three glasses of non-caffeinated beverages prior to arrival to facilitate the collection of a baseline urine collection and an additional two to five glasses upon arrival at the CTRC.

Upon arrival on the morning of the study visit, the nursing staff will ask the study subject to provide verbal confirmation that they took the KI pill and will document and record on the study flow sheet the approximate time that the subject took the tablet. If the pill was not taken within the allowed time range of 6:00 AM to 10:00 AM, the subject will not be able to participate in the study visit. A research team member will obtain informed consent from the participant and a copy of the consent will be given to the subject. The nursing staff will measure and record the subject's height, weight, blood pressure, temperature, pulse rate, respiration rate; confirm that the subject has not experienced any changes in physical/psychological health since the screening; and collect a baseline urine sample. As outlined above, if three weeks or more has elapsed since the health screening, women of childbearing age will be administered a urine pregnancy test, prior to the insertion of the IV lines, using an aliquot of the baseline urine sample. The test kits used will be purchased from a local pharmacy by the site principal investigator or her delegate and provided to the CTRC staff. Nursing will interpret the results of the test and the principal investigator will verify a negative result prior to initiation of the GFR measurement. If the test yields a positive result, the study visit will be immediately terminated.

Subjects with diabetes will be requested to bring their own testing devices. The CTRC has their own testing devices if the subject forgets to bring his or her own. Subjects will be asked to check their blood sugar upon arrival at the CTRC. If they are unable to perform the measurement, the nurses will do so. The study physician will be informed of low (less 100 mg/dl) or high (greater than 200) blood sugars. Otherwise, the participant will follow their normal routine for checking blood sugar. For example, if they check after each meal, then they will be asked to do so. If they only check once a day, then they will not be asked to check again. Participants will be fed breakfast and lunch and therefore there is no concern for hypoglycemia over the course of the study visit.

A saline lock and intravenous line will be inserted at two different sites and two drops of saturated solution of potassium iodide (SSKI) will be administered at least 30 minutes and no more than six hours prior to the administration of 125I-iothalamate to prevent uptake by the thyroid. Baseline laboratory tests will include serum creatinine, cystatin C, blood urea nitrogen (BUN), C-reactive protein (CRP), electrolytes and albumin.

The markers to be administered will be prepared by a pharmacist at the Tufts Medical Center Pharmacy. The pharmacist will prepare the markers such that they can be administered directly by the nurse. That is, the correct dose will be placed in a syringe that can be administered directly to the participant. A member of the research team will obtain the drugs and bring them to the CTRC for administration by the nurse.

After collection of the baseline blood sample and a separate sample for tissue banking (optional), 50 mg Inulin/kg will be administered by bolus IV, followed by a sustaining dose of 18.8 mg/square area/min. Approximately 30 minutes later, 35 µCuries of 125I-iothalamate will be injected subcutaneously to allow for a 60 minute equilibrium time. After a further 30 minutes, 5 ml of Iohexol (Omnipaque 300, 300mg/mL of organic iodine) and 10 uL/kg of Gd-DTPA will be administered via a bolus IV injection through the same IV line as inulin. Iohexol will be given first over 1 minute, followed by saline flush of the intravenous line, followed by Gd-DTPA over one minute. Subjects with an eGFR < 30 mL/min/1.73 m2, as determined from their medical record or the serum creatinine measurement from the health screening, will not receive Gd-DTPA. The syringes used to administer the iohexol and Gd-DTPA will be weighed to the nearest tenth gram on the same scale before and after injection. Nurses at the CTRC will monitor the participant at the time of the administration and throughout the study.

Blood samples for plasma clearance measurements will be obtained from the second IV line, which will also remain in place throughout the course of the study visit. To maintain the patency of the IV access for the purpose of the serial blood collections, normal saline will be administered at a rate of approximately 20-30 c.c. per hour from a 500 c.c. bag of normal saline.

The administration of inulin will be considered time 0. Following the iohexol administration, blood samples will be taken at approximately 10, 30, 120, and 240 minutes from the second intravenous line. For participants with estimated GFR less than 45 ml/min per 1.73 m2, as determined from the screening visit or the subject's medical record, a sample will be drawn at 360 minutes. The exact time of the sample will be recorded.

Following the 180-minute timed void, all voluntary voids will be collected but the volume of oral fluid intake will match the urine output (i.e. water loading to stop). The nursing staff will continue to monitor fluid balance. For all urine samples, a bladder scan will be conducted immediately before and immediately after the subject urinates to assess the completeness of bladder emptying. Following the equilibration period for inulin (90 minutes) and 125I-iothalamate (60 minutes), four timed urinary clearance periods of at least 30 minutes will begin. Blood samples for urinary clearance measurements will be taken following each bladder emptying. Blood samples for plasma clearance measurements will be taken at approximately 10, 30, 120, 150, and 240 min. For patients with estimated GFR <30 mL/min per 1.73 m2, an additional blood sample will be collected at 360 min. Subjects are free to move around during the GFR test.

Participants will be fed a breakfast consisting of a standardized protein content following collection of the 30 minute blood sample and a lunch of similar protein content. Subjects with diabetes will be given a meal that is consistent with their treatment regimen and asked to administer their medications and check their blood sugar levels during the course of the study visit as they would normally do, in the manner prescribed by their treating physician.

At the conclusion of the study, both intravenous lines will be removed. Subjects will remain at the CTRC for at least 30 minutes following removal of the IV lines. During that time, nursing staff will re-measure and record the subject's vital signs (height, weight, blood pressure, temperature, pulse rate, respiration rate). Upon successful completion of a study visit, subjects will receive a stipend

Subjects will undergo repeat study visits with a target time of one month between visits. The second study visit will proceed in an identical manner with the exception that urinary clearance of inulin will only be measured in a subset of the study participants during the second visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Older than 18 years of age.
* With and without known CKD - for the purpose of this study, CKD will be defined on the basis by prior diagnosis of CKD, urologic or kidney disease, known abnormal urinalysis, or history of having seen a nephrologist.

Exclusion Criteria:

* Currently undergoing or having received peritoneal dialysis or hemodialysis treatment within the past three months. Subjects with an eGFR < 30 mL/min/1.73 m2 will not receive Magnevist during the study visit.
* Active pulmonary edema.
* Class III or IV congestive heart failure.
* History of urinary retention or current urinary incontinence.
* Inability to cease taking medications that affect creatinine levels (e.g., bactrim, cimetidine) for one week prior to the study visit.
* Inability to maintain a stable regimen of anti-inflammatory agents and angiotensin converting enzyme inhibitors for one week prior to study visit
* Current treatment with amiodarone or metformin.
* Acute exacerbation of asthma or chronic obstructive lung disease in the past three months requiring hospitalization or oral steroid therapy.
* Inadequate venous access.
* End stage conditions such as cirrhosis.
* Active treatment for cancer.
* Progressive neurological diseases.
* Severe gastric immotility.
* Recent radiation exposure to γ-emitting isotope other than technetium
* Known allergy to any of the GFR markers, iodine, or shellfish. Subjects who are not sure if they have an iodine allergy because they have not eaten shellfish or have never received contrast dye will be excluded from participation.
* Dermatitis herpetiformis.
* Hypocomplementemic vasculitis.
* Multinodal goiter.
* Graves' disease.
* Autoimmune thyroiditis.
* Cognitive or physical impairments that will prevent a subject from providing informed consent.
* History of mastectomy.
* Hemoglobin levels below 10 g/dL.
* Women who are either pregnant or who intend to become pregnant during the period of time in which the study visits will occur.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with CKD and without CKD will be recruited to participate in the study. Subjects with CKD will be recruited primarily from the Kidney and Blood Pressure Center. Subjects without CKD will be recruited from advertisements as well as the volunteer database at the Jean Mayer Human Nutrition Research Center on Aging (HRNCA), which is located next to Tufts Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Accuracy and precision of the different markers for measuring GFR | End points are not applicable. It's a cross-sectional design study

CONTACTS AND LOCATIONS:
Overall Officials: Lesley A Stevens, MD, MS, Principal Investigator — Tufts Medical Center